CLINICAL TRIAL: NCT05811247
Title: Phase 3 Randomized Double-Blind Placebo-Controlled 1-year Parallel-Arm Study to Compare a Fixed Dose Combination of Aroxybutynin/Atomoxetine (AD109) to Placebo in Obstructive Sleep Apnea (LunAIRo Study)
Brief Title: Parallel Arm Trial of AD109 and Placebo With Patients With OSA (LunAIRo)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Apnimed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APC-APN-304
Record Dates: First submitted 2023-03-31; First posted 2023-04-13 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: OSA
Keywords: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AD109 (Experimental): AD109
  Interventions: Drug: AD109
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AD109 — Oral administration at bedtime.
  Arms: AD109
Drug: Placebo — Oral administration at bedtime.
  Arms: Placebo

SUMMARY:
This is a Phase 3 Randomized Double-Blind Placebo-Controlled 1-year Parallel-Arm Study to Compare a Fixed Dose Combination of AD109 to Placebo in Obstructive Sleep Apnea.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age at the time of informed consent.
2. PSG criteria: AHI of >5; ≤ 25% central or mixed apneas; and PLM arousal index ≤15
3. PROMIS-Fatigue: raw score ≥17
4. PAP intolerance or current PAP refusal.
5. BMI between 18.5 and 40 kg/m2 for men, or 42 kg/m2 for women, inclusive.

Exclusion Criteria:

1. Narcolepsy, restless leg syndrome, REM sleep behavior disorder
2. Insomnia disorder characterized by difficulty initiating or maintaining sleep, or use within the past month of sedative-hypnotics or other medication for the purpose of treating or avoiding insomnia symptoms.
3. Pierre Robin, Treacher Collins, or other craniofacial malformation syndrome, or grade ≥3 tonsillar hypertrophy.
4. Clinically significant cardiac disease, e.g., ventricular arrhythmia, untreated or unstable coronary artery disease, cardiac failure. Stable atrial arrhythmia is allowed.
5. Neuromuscular disorder (e.g., motor neuron disease, muscular dystrophy or myopathy, myasthenic syndrome); epilepsy; Parkinson, Alzheimer, or other neurodegenerative disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660 (Actual)
Dates: Start 2023-08-28 (Actual); Primary Completion 2025-05-07 (Actual); Study Completion 2025-05-07 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Apnea-Hypopnea Index (AHI) | 6 months
  AHI, Apnea-Hypopnea Index, is the number of apneas or hypopneas recorded via polysomnography during the study per hour of sleep. Apnea is defined as a cessation of airflow lasting at least 10 seconds, hypopnea as a decrease in airflow by at least 30% from baseline for at least 10 seconds occurring with a drop in oxygen saturation (SpO2) by at least 4%.

CONTACTS AND LOCATIONS:
Locations (64):
- United States (64):
  - Sleep Disorders Center of Alabama, Birmingham, Alabama
  - Chandler Clinical Trials, Chandler, Arizona
  - Preferred Research Partners, Inc., Little Rock, Arkansas
  - Orange County Research Institute, Anaheim, California
  - Marvel Clinical Research, LLC, Huntington Beach, California
  - CenExel CNS, Los Alamitos, California
  - Santa Monica Clinical Trials, Los Angeles, California
  - Empire Clinical Research, Pomona, California
  - Pacific Research Network, San Diego, California
  - SDS Clinical Trials Inc., Santa Ana, California
  - Alpine Clinical Research Center, Boulder, Colorado
  - Mountain View Clinical Research, Inc., Denver, Colorado
  - Nuvance Health, Norwalk, Connecticut
  - Teradan Clinical trials LLC, Brandon, Florida
  - St. Francis Medical Institute, Clearwater, Florida
  - Nouvelle Clinical Research, Cutler Bay, Florida
  - Arrow Clinical Trials, Daytona Beach, Florida
  - Cenexel Research Centers of America - Hollywood, Hollywood, Florida
  - Ivetmar Medical Group LLC, Miami, Florida
  - PharmaDev Clinical Research Institute, LLC, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Palm Beach Research ClinEdge-PPDS, West Palm Beach, Florida
  - Clinical Site Partners, LLC dba Flourish Research, Winter Park, Florida
  - NeuroTrials Research, Atlanta, Georgia
  - CenExel iResearch, Decatur, Georgia
  - Sleep Practitioners, LLC, Macon, Georgia
  - Centricity Research Rincon Pulmonology, Rincon, Georgia
  - Medster Research, Valdosta, Georgia
  - Chicago Research Center Inc, Chicago, Illinois
  - Sleep Disorders Centers of the Mid-Atlantic, Glen Burnie, Maryland
  - Velocity Clinical Research, Rockville, Maryland
  - Neurocare, Inc, Newton, Massachusetts
  - Infinity Medical Research, North Dartmouth, Massachusetts
  - Baystate Medical Center (BMC) - Baystate Sleep Medicine, Springfield, Massachusetts
  - Western Michigan University Homer Stryker M.D. School of Medicine, Kalamazoo, Michigan
  - Henry Ford Health (Sleep Research Department), Novi, Michigan
  - Clinical Neurophysiology Services, Sterling Heights, Michigan
  - St Lukes Hospital, Chesterfield, Missouri
  - Healthcare Research Network, Hazelwood, Missouri
  - Clayton Sleep Institute, St Louis, Missouri
  - Great Plains Health, North Platte, Nebraska
  - Henderson Clinical Trials, Henderson, Nevada
  - Clinilabs, Inc, Eatontown, New Jersey
  - Maimonides Sleep Arts and Sciences, Albuquerque, New Mexico
  - Northwell Health Physician Partners, New Hyde Park, New York
  - Research Carolina Elite, Denver, North Carolina
  - Clinical Research of Gastonia, Gastonia, North Carolina
  - Advanced Respiratory and Sleep Medicine, LLC, Huntersville, North Carolina
  - Coastal Carolina Health Care, New Bern, North Carolina
  - Meridian Clinical Research, Raleigh, North Carolina
  - NeuroScience Research Center, LLC, Canton, Ohio
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Sleep Management Institute, Cincinnati, Ohio
  - Ohio Sleep Medicine Institute, Dublin, Ohio
  - Northwest Research Center, Portland, Oregon
  - Brian Abaluck, LLC, Malvern, Pennsylvania
  - UPMC Comprehensive Lung Center - Sleep Medicine, Pittsburgh, Pennsylvania
  - Lowcountry Lung and Critical Care, Charleston, South Carolina
  - Velocity Clinical Research - Greenville, Greenville, South Carolina
  - Clinical Neuroscience Solutions - Memphis, Memphis, Tennessee
  - FutureSearch Trials of Neurology, Austin, Texas
  - Central Texas Neurology Consultants, PA, Round Rock, Texas
  - Sleep Therapy Research Center, San Antonio, Texas
  - Sleep Disorders Centers of the Mid-Atlantic, Vienna, Virginia